CLINICAL TRIAL: NCT03167073
Title: Impact of a Novel Smartphone Application on Postpartum Weight Loss and Breastfeeding Rates Among Low-income, Urban Women
Brief Title: Impact of a Smartphone Application on Postpartum Weight Loss and Breastfeeding Rates Among Low-income, Urban Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 201704147
Record Dates: First submitted 2017-05-15; First posted 2017-05-25 (Actual); Results first posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Breastfeeding
Keywords: smartphone application; low-income women; breastfeeding; health education; health disparities; postpartum weight loss
MeSH Terms: conditions — Breast Feeding; Health Education

STUDY DESIGN:
Intervention Model Description: All participants will receive a complementary android phone with 3 months of complementary internet service upon enrollment at approximately 36 weeks gestation. Women will be randomized to receiving Breastfeeding Friend (BFF; the intervention) or a dummy app (control), which looks identical to BFF but contains limited breastfeeding content available during routine prenatal care.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The coding team has labeled BFF and the dummy app as "BFF-1" and BFF-2." The research team is blinded to which app is BFF-1 and which is BFF-2. Sprint Telecommunications will receive the .apks files for both apps and load one app to each research phone according to the randomization algorithm that researchers at Washington University will provide to them. This algorithm has been created to randomize participants in blocks of four. Sprint will then send the phones to the research team with labels on the box that state the research phone number and app number (ie, phone 18, BFF-2). Participants will be given the phones in a sequential manner. After the study is completed, the researchers will contact the coding team, and the study will be un-blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BreastFeeding Friend (BFF) (Experimental): BFF is a novel android app initially created in Microsoft PowerPoint with the results of a well-validated questionnaire administered to the target patient population, in which participants identified barriers preventing them from starting or continuing breastfeeding. The app was then modified by a multidisciplinary team of neonatologists, perinatologists, and certified lactation consultants. The finalized prototype was presented to three focus groups of test users sociodemographically similar to the target population. This approach allowed BFF to be adjusted to maximize the users' experience per their opinions. Once the focus groups' feedback was consistent, the app prototype was provided to a freelance coding team at Washington University of St. Louis, which built a native android app.
  Interventions: Other: BreastFeeding Friend (BFF)
- dummy app (Placebo Comparator): The dummy app looks identical to BFF but is limited to a few pages of information on breastfeeding that is provided in hand-out form during routine prenatal care.
  Interventions: Other: dummy app

INTERVENTIONS:
Other: BreastFeeding Friend (BFF) — A novel android app designed to improve breastfeeding rates among low-income women
  Arms: BreastFeeding Friend (BFF)
Other: dummy app — A novel android app that looks identical to the intervention app (BFF) but contains limited content.
  Arms: dummy app

SUMMARY:
Breastfed babies have significant health benefits extending beyond infancy, including lower rates of childhood obesity and infection. Mothers who breastfeeding also have health benefits, including increased rates of postpartum weight loss. Low-income women are less likely to breastfeed comparatively; this disparity may be due to misconceptions about breastfeeding benefits or poor social support. Based on survey results and focus groups of low-income women, the investigators designed a novel smart-phone application to confront barriers women perceived prevented them from breastfeeding and propose the first-ever randomized controlled trial describing the impact a smart phone app has on postpartum weight loss and breastfeeding rates among low-income women.

DETAILED DESCRIPTION:
Breastfed babies have fewer childhood infections than formula-fed babies, and women who breastfeed have a reduced risk of cardiovascular disease and increased rates of postpartum weight loss. Thus, the American College of Obstetricians and Gynecologists (ACOG) recommends six months of exclusive breastfeeding after birth. Nationally, 75% of women initiate breastfeeding, but only 59% of Black women, 53% of teenagers, and 66% of women in the Special Supplemental Nutrition Program for Women, Infants, and Children breastfeed. Unpublished internal data suggest that, while the breastfeeding initiation rate for women receiving prenatal care at Barnes-Jewish Hospital's Medicaid clinic is higher than the national average (89%), by postpartum day #2, only 34% exclusively breastfeed. Reasons for this precipitous decline in breastfeeding are not fully understood but include misconceptions about breastfeeding benefits and poor social support.

This study would be the first-ever randomized controlled trial describing the impact that a smart phone application (app) has on breastfeeding rates and thus postpartum weight loss among low-income women. In this study's first phase, a previously well-validated questionnaire was used to identify barriers that low-income urban women perceived as preventing breastfeeding initiation or continuation. In the second phase, these data-as well as input from neonatologists, certified lactation consultants, and focus groups of low-income pregnant women-were used to create a smart phone application (app) to promote breastfeeding called Breastfeeding Friend (BFF). The investigators chose an app to provide breastfeeding support for two reasons. First, nearly two-thirds of American adults, and 90% of those under the age of 29, have smart phones. Second, more than two-thirds of Americans with smart phones use them to obtain health information via new media (blogs, websites, and apps). Among low-income women, physician-designed new media have improved intrauterine device uptake rates and decreased rates of postpartum smoking. BFF will serve as a virtual lactation consultant, increasing breastfeeding knowledge while providing interactive assistance and access to in-person resources. By providing women with more breastfeeding support, this app could increase postpartum weight loss by decreasing a significant health disparity.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous women with non-anomalous singleton pregnancies who speak English and do not have contraindication for breastfeeding. They must receive prenatal care at the Washington University in St. Louis's Center for Outpatient Health, the Medicaid clinic. Recruitment will occur at around 36 weeks gestation.

Exclusion Criteria:

* multiparous women with contraindications to breastfeeding, multiple gestations, an anomalous fetus, or who do not speak English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must be pregnant to participate.
Enrollment: 170 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam K Lewkowitz, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Center for Outpatient Health, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided
Once unblinded, the investigators may elect to make all de-identified IPD available to other researchers.

REFERENCES:
- [Derived] Griffin LB, Lopez JD, Ranney ML, Macones GA, Cahill AG, Lewkowitz AK. Effect of Novel Breastfeeding Smartphone Applications on Breastfeeding Rates. Breastfeed Med. 2021 Aug;16(8):614-623. doi: 10.1089/bfm.2021.0012. Epub 2021 Apr 7. PMID 33826418
- [Derived] Lewkowitz AK, Lopez JD, Carter EB, Duckham H, Strickland T, Macones GA, Cahill AG. Impact of a novel smartphone application on low-income, first-time mothers' breastfeeding rates: a randomized controlled trial. Am J Obstet Gynecol MFM. 2020 Aug;2(3):100143. doi: 10.1016/j.ajogmf.2020.100143. Epub 2020 May 17. PMID 33345878
- [Derived] Lewkowitz AK, Lopez JD, Werner EF, Ranney ML, Macones GA, Rouse DJ, Savitz DA, Cahill AG. Effect of a Novel Smartphone Application on Breastfeeding Rates Among Low-Income, First-Time Mothers Intending to Exclusively Breastfeed: Secondary Analysis of a Randomized Controlled Trial. Breastfeed Med. 2021 Jan;16(1):59-67. doi: 10.1089/bfm.2020.0240. Epub 2020 Oct 20. PMID 33085510

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BreastFeeding Friend (BFF) | Dummy App
Started | 85 | 85
Completed | 84 | 85
Not Completed | 1 | 0
Not completed — Stillbirth | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BreastFeeding Friend (BFF) | Dummy App | Total
Number analyzed (Participants) | 84 | 85 | 169
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 8 | 19
  Between 18 and 65 years | 73 | 77 | 150
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.7 (4.9) | 21.6 (4.0) | 22.2 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 85 | 169
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 83 | 83 | 166
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 71 | 67 | 138
  White | 9 | 10 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  United States | 84 | 85 | 169

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Breastfeeding Without Formula Supplementation
Description: Number of participants breastfeeding without formula supplementation. This was obtained via confidential questionnaire
Time Frame: Postpartum day number 2
Measure: Count of Participants; unit: Participants
Arm/Group | BreastFeeding Friend (BFF) | Dummy App
Number analyzed (Participants) | 84 | 85
Participants | 30 | 30

2. Secondary Outcome: Postpartum Weight Loss
Description: Postpartum weight loss will be measured by subtracting reported weight at postpartum month 6 obtained from confidential postpartum month 6 survey from measured weight obtained in-person at hospital on postpartum day 2
Time Frame: Participants will be weighed in-person on postpartum day 2. Survey at postpartum month 6 will prompt participant to weigh herself and include this weight on the survey.
Population: Data were not collected for this outcome because owning a home scale was not a requirement for study eligibility, and women in our study population did not own scales at home so were unable to provide weights at 6 months postpartum.
Arm/Group | BreastFeeding Friend (BFF) | Dummy App
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants Breastfeeding Without Formula Supplementation
Description: Number of participants breastfeeding without formula supplementation; to be obtained via confidential questionnaire
Time Frame: postpartum week 6
Population: Data were missing from 1 participant in the BFF group. Participants with missing data were excluded from analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | BreastFeeding Friend (BFF) | Dummy App
Number analyzed (Participants) | 83 | 85
Participants | 12 | 14

4. Secondary Outcome: Number of Participants Breastfeeding Without Formula Supplementation
Description: Number of participants breastfeeding without formula supplementation, to be obtained via confidential questionnaire
Time Frame: postpartum month 3
Population: Data were missing from 8 participants in the BFF group and 9 participants in the dummy app group. Participants with missing data were excluded from analysis for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | BreastFeeding Friend (BFF) | Dummy App
Number analyzed (Participants) | 76 | 76
Participants | 10 | 10

5. Secondary Outcome: Number of Participants Breastfeeding Without Formula Supplementation
Description: Number of participants breastfeeding without formula supplementation; to be obtained via confidential questionnaire
Time Frame: postpartum month 6
Population: Data were missing from 24 participants in the BFF group and 18 participants in the dummy app group. Participants with missing data were excluded from analysis for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | BreastFeeding Friend (BFF) | Dummy App
Number analyzed (Participants) | 60 | 67
Participants | 5 | 7

6. Secondary Outcome: Number of Participants Breastfeeding With or Without Formula Supplementation
Description: Number of participants breastfeeding with or without formula supplementation; to be obtained via confidential questionnaire
Time Frame: postpartum day 2
Measure: Count of Participants; unit: Participants
Arm/Group | BreastFeeding Friend (BFF) | Dummy App
Number analyzed (Participants) | 84 | 85
Participants | 62 | 66

7. Secondary Outcome: Number of Participants Breastfeeding With or Without Formula Supplementation
Description: as for outcome 6
Time Frame: postpartum week 6
Population: Data were missing from 1 participants in the BFF group. Participants with missing data were excluded from analysis for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | BreastFeeding Friend (BFF) | Dummy App
Number analyzed (Participants) | 83 | 85
Participants | 39 | 49

8. Secondary Outcome: Number of Participants Breastfeeding With or Without Formula Supplementation
Description: as for outcome 6
Time Frame: postpartum month 3
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | BreastFeeding Friend (BFF) | Dummy App
Number analyzed (Participants) | 76 | 76
Participants | 23 | 28

9. Secondary Outcome: Number of Participants Breastfeeding With or Without Formula Supplementation
Description: as for outcome 6
Time Frame: postpartum month 6
Measure: Count of Participants; unit: Participants
Arm/Group | BreastFeeding Friend (BFF) | Dummy App
Number analyzed (Participants) | 60 | 67
Participants | 10 | 16

10. Other Pre Specified Outcome: Number of Participants Reporting That App is Best Breastfeeding Resource
Description: App is best breastfeeding resource, measured by confidential questionnaire
Time Frame: postpartum week 6
Population: Data were missing from 19 participants in the BFF group and 21 participants in the dummy app group. Participants with missing data were excluded from analysis for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | BreastFeeding Friend (BFF) | Dummy App
Number analyzed (Participants) | 65 | 64
Participants | 34 | 20

ADVERSE EVENTS:
Time Frame: From enrollment until study completion (7 months per participant). 2 year study dureation.
Description: Same as clinicaltrial.gov definitions
Arm/Group | BreastFeeding Friend (BFF) | Dummy App
All-Cause Mortality (participants affected / at risk) | 0/84 | 0/85
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/85
Other Adverse Events (participants affected / at risk) | 0/84 | 0/85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT03167073/Prot_SAP_000.pdf